CLINICAL TRIAL: NCT01593345
Title: Promotion of Self-management of Chronic Mobility Limitations Among Vulnerable Seniors at the MUHC: Training the New Generation of Canadian Physiotherapists for This Role. Addendum: Planning Physiotherapy Services for Persons Treated at the MUHC for Cancer: A Needs Assessment
Brief Title: Self-management of Chronic Mobility Limitations in MUHC Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Richard and Edith Strauss Foundation of Canada (Unknown)
Responsible Party: Principal Investigator, Nancy Mayo, Dr, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2476
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Seniors With Mobility Limitations
Keywords: Elderly; mobility limitations; self-management; exercise
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mentor (Experimental)
  Interventions: Other: Mobility self-management with Mentor
- Guidebook (Active Comparator)
  Interventions: Other: Mobility self-management with guidebook

INTERVENTIONS:
Other: Mobility self-management with Mentor — will be offered an evaluation and treatment plan supervised by a qualified physiotherapist, accompanied by written and visual material to enhance mobility self-management skills, supported by telephone mentoring by physiotherapy students in the Professional Master's program. The components of the mobility self-management program will target skill enhancement of each senior to identify their functional limitations, set realistic goals for mobility improvement, develop a mobility action plan, carry out the plan, and then re-assess their function and mobility. Mobility self-assessment, personalized goals, and the action plan will be incorporated into a personalized workbook that the senior can use to monitor their function profile and serve as a communication aid during health care encounters.
  Arms: Mentor
Other: Mobility self-management with guidebook — will be mailed an exercise guide targeting the key mobility limitations common in the elderly (range of motion, arm, leg, and core strength, and breathing). This guide has been developed and has been pilot tested on a small number of seniors and has been shown to be acceptable and feasible.
  Arms: Guidebook

SUMMARY:
The population is aging and chronic conditions, which are major causes of pain and mobility limitations, are on the rise, however, current access to physiotherapy is difficult. Knowledge on managing disability is substantial, but methods to translate into action are lacking. This project is designed to test a novel method of promoting function in vulnerable seniors and simultaneously develop awareness in the new generation of physiotherapists that they can have a proactive role in health promotion. The investigators are proposing a pilot project targeting both students and patients.

The research question are (1) What are the needs of vulnerable patients at the MUHC? Two groups will be targeted; newly discharged seniors (who will be eligible for an intervention) and cancer outpatients who will be surveyed only);(2) For a senior population at risk for physical deterioration, to what extent is a personalized mentoring approach to optimizing function and preventing disability through developing self-management skills more effective in improving outcomes than the provision of written material covering the same general content? (3) Does a mentoring experience with vulnerable seniors through development and teaching of a self-management program (comprised of education and support) produce meaningful positive changes in future clinicians' knowledge, skills and attitude towards modes of delivering physiotherapy services and promoting self-management in Canadian seniors?

There are two phases to this study: a survey and randomized controlled trial (RCT). The survey phase will identify mobility needs of two groups, newly discharged seniors and cancer outpatients. The needs assessment for newly discharged seniors will identify people eligible for the (RCT) component; the needs assessment for cancer outpatients will inform the development of interventions for this specific group. The RCT component will be piloted for recently discharged community dwelling seniors 70 years and older only.

A sample of 400 seniors recently discharged from the adult, general, hospital sites of the MUHC will be contacted for a needs assessment. From this pool, the investigators anticipate 100 will be eligible and 60 will be randomized, 30 to the mentor intervention and 30 to the control group. Participants will be followed-up for 6 months and assessments will be performed at 2 time points (baseline and 6 months). The main outcome is a standardized response ratio (SRR) estimated across all persons and measures. SRRs will be calculated for three groups of response variables: impairment/mobility measures, quality of life indicators, and health services outcomes.

In parallel, to determine cancer survivor needs, the investigators will contact 600 cancer survivors; as the investigators anticipate 400 will answer the survey. The analysis of this survey will consist of frequency of specific needs by diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* community dwelling seniors,
* aged 70 years and older,
* recently discharged from one of the adult general (MGH, RVH, Lachine) hospital sites,
* with anyone of the following mobility limitations:

  1. Limitation in walking more than 1 block
  2. Limitation in going up 1 flight of stairs
  3. Unable to get groceries without help
  4. Unable to do housework (dishes, meals, vacuuming, making bed) without help
  5. Self-rated health fair or poor
  6. Pain
  7. Shortness of breath

Exclusion Criteria:

* seniors discharged with orthopaedic or cardiac surgery, or
* with stroke or myocardial infarction, as formal rehabilitation is part of the usual care plan for these conditions.

Also excluded will be people with dementia as identified on the medical chart.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Brief Pain Questionnaire | 2 time points (baseline and 6 months)
DASH | 2 time points (baseline and 6 months)
LEFS | 2 time points (baseline and 6 months)
RAND-MOS36 | 2 time points (baseline and 6 months)
Short Self Efficacy scale | 2 time points (baseline and 6 months)

SECONDARY OUTCOMES:
Health care utilization | 2 time points (baseline and 6 months)
Medication management | 2 time points (baseline and 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Mayo, PhD, Principal Investigator — McGill University
Locations (3):
- Canada (3):
  - Lachine Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Background] Raina P, Dukeshire S, Lindsay J, Chambers LW. Chronic conditions and disabilities among seniors: an analysis of population-based health and activity limitation surveys. Ann Epidemiol. 1998 Aug;8(6):402-9. doi: 10.1016/s1047-2797(98)00006-4. PMID 9708876
- [Background] Passalent LA, Landry MD, Cott CA. Exploring wait list prioritization and management strategies for publicly funded ambulatory rehabilitation services in ontario, Canada: further evidence of barriers to access for people with chronic disease. Healthc Policy. 2010 May;5(4):e139-56. PMID 21532763
- [Background] Marks R, Allegrante JP, Lorig K. A review and synthesis of research evidence for self-efficacy-enhancing interventions for reducing chronic disability: implications for health education practice (part I). Health Promot Pract. 2005 Jan;6(1):37-43. doi: 10.1177/1524839904266790. PMID 15574526
- [Background] Marks R, Allegrante JP, Lorig K. A review and synthesis of research evidence for self-efficacy-enhancing interventions for reducing chronic disability: implications for health education practice (part II). Health Promot Pract. 2005 Apr;6(2):148-56. doi: 10.1177/1524839904266792. PMID 15855284
- [Background] Daniels R, van Rossum E, de Witte L, Kempen GI, van den Heuvel W. Interventions to prevent disability in frail community-dwelling elderly: a systematic review. BMC Health Serv Res. 2008 Dec 30;8:278. doi: 10.1186/1472-6963-8-278. PMID 19115992
- [Background] Fritz JM, Hunter SJ, Tracy DM, Brennan GP. Utilization and clinical outcomes of outpatient physical therapy for medicare beneficiaries with musculoskeletal conditions. Phys Ther. 2011 Mar;91(3):330-45. doi: 10.2522/ptj.20090290. Epub 2011 Jan 13. PMID 21233306
- [Background] Graham ID, Logan J, Harrison MB, Straus SE, Tetroe J, Caswell W, Robinson N. Lost in knowledge translation: time for a map? J Contin Educ Health Prof. 2006 Winter;26(1):13-24. doi: 10.1002/chp.47. PMID 16557505
- [Background] Wagner EH, Davis C, Schaefer J, Von Korff M, Austin B. A survey of leading chronic disease management programs: are they consistent with the literature? Manag Care Q. 1999 Summer;7(3):56-66. PMID 10620960
- [Background] Wagner EH, Austin BT, Davis C, Hindmarsh M, Schaefer J, Bonomi A. Improving chronic illness care: translating evidence into action. Health Aff (Millwood). 2001 Nov-Dec;20(6):64-78. doi: 10.1377/hlthaff.20.6.64. PMID 11816692
- [Background] Chodosh J, Morton SC, Mojica W, Maglione M, Suttorp MJ, Hilton L, Rhodes S, Shekelle P. Meta-analysis: chronic disease self-management programs for older adults. Ann Intern Med. 2005 Sep 20;143(6):427-38. doi: 10.7326/0003-4819-143-6-200509200-00007. PMID 16172441
- [Background] Kennedy A, Reeves D, Bower P, Lee V, Middleton E, Richardson G, Gardner C, Gately C, Rogers A. The effectiveness and cost effectiveness of a national lay-led self care support programme for patients with long-term conditions: a pragmatic randomised controlled trial. J Epidemiol Community Health. 2007 Mar;61(3):254-61. doi: 10.1136/jech.2006.053538. PMID 17325405
- [Background] Kennedy A, Rogers A, Bower P. Support for self care for patients with chronic disease. BMJ. 2007 Nov 10;335(7627):968-70. doi: 10.1136/bmj.39372.540903.94. PMID 17991978
- [Background] King AC, Pruitt LA, Phillips W, Oka R, Rodenburg A, Haskell WL. Comparative effects of two physical activity programs on measured and perceived physical functioning and other health-related quality of life outcomes in older adults. J Gerontol A Biol Sci Med Sci. 2000 Feb;55(2):M74-83. doi: 10.1093/gerona/55.2.m74. PMID 10737689
- [Background] Lazowski DA, Ecclestone NA, Myers AM, Paterson DH, Tudor-Locke C, Fitzgerald C, Jones G, Shima N, Cunningham DA. A randomized outcome evaluation of group exercise programs in long-term care institutions. J Gerontol A Biol Sci Med Sci. 1999 Dec;54(12):M621-8. doi: 10.1093/gerona/54.12.m621. PMID 10647968
- [Background] Kramer AF, Erickson KI, Colcombe SJ. Exercise, cognition, and the aging brain. J Appl Physiol (1985). 2006 Oct;101(4):1237-42. doi: 10.1152/japplphysiol.00500.2006. Epub 2006 Jun 15. PMID 16778001
- See also: Portrait of Seniors in Canada. — http://www.statcan.gc.ca/pub/89-519-x/89-519-x2006001-eng.pdf
- See also: Percentage of persons who are active, moderately active or inactive, by age group. — http://www.statcan.gc.ca/pub/89-519-x/2006001/t/4181621-eng.htm